CLINICAL TRIAL: NCT05972837
Title: Effects of Home-based Surface Electrical Stimulation for Patients with Cervical Myofascial Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Director of Physical Medicine and Rehabilitation, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202204099
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Myofascial Pain Syndrome of Neck
Keywords: Myofascial Pain Syndromes; Surface electrical stimulation; Remote medical support; Telemedicine
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SES combined with telemedical support (Experimental): SES device for personal use will be provided for participants in addition to remote medical support.
  Interventions: Device: Surface electrical stimulation (SES); Other: Remote medical support
- SES (Active Comparator): Participants in this group will also attend an appointment via a video call with a rehabilitation doctor in the first week but no weekly telehealth visits. Only SES device for personal use and a user manual will be provided.
  Interventions: Device: Surface electrical stimulation (SES)
- No intervention (No Intervention): Participants in this group will not be provided either SES device or weekly telehealth visits. They are only required to attend a session of video call with a rehabilitation doctor in the first week.

INTERVENTIONS:
Device: Surface electrical stimulation (SES) — Participants will undergo 3 weeks (20 minutes/ time, three times/ week) of SES intervention.
  Arms: SES; SES combined with telemedical support
Other: Remote medical support — The remote medical support includes a session of video call with a rehabilitation doctor in the first week and weekly telehealth visits with a live physical therapist or physician. The contents of the video calls contain patient education, stretching exercises teaching and instructions of using SES for MPS.
  Arms: SES combined with telemedical support

SUMMARY:
The aim of this study is to compare the developed home-based surface electrical stimulation program to the controls in computer office workers with MPS.

DETAILED DESCRIPTION:
Cervical myofascial pain syndrome (MPS) is a common problem among workers who have large amount of computer use. Additionally, owing to the high workload and long hours of staying in thier cubicle, the office employees are often unable to have extra time to receive rehabilitation and treatment regularly. A home-based surface electrical stimulation (SES) program is developed to help intervention be time-saving and more accessible for office-based staff busy at work.

In this single-blind randomized controlled trial, participants will be assigned to one of the following three groups and undergo 3 weeks (20 minutes/ time, three times/ week) of intervention:

1. SES combined with telemedical support
2. SES
3. No intervention

The outcome assessments will be performed before and after the intervention (0-wk and 4-wk) and 4 weeks after the endpoint of intervention (8-wk). The outcome assessor was blind to the intervention and group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Time of using computer > 4hrs/day
* Neck pain > 2 months
* Diagnosis of cervical myofascial pain syndrome
* VAS pain ≥ 3 (0~10)

Exclusion Criteria:

* Had a history of neck surgery
* Pregnancy
* Systematic disease (e.g. autoimmune disorders, arthritis, infection, etc.)
* Malignancy
* Neurological signs such as radiating pain, motor weakness in the upper extremities.
* Skin defect or scars at the planned placement of SES
* Pacemaker user
* History of seizure attack
* History of diabetes
* Fear of receiving SES

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  A visual analog scale (VAS, scoring from 0-10) is used to measure a participant's pain intensity. The participant indicates their level of pain on average over the past 3 days.

SECONDARY OUTCOMES:
Pain intensity | 8 weeks
  A visual analog scale (VAS, scoring from 0-10) is used to measure a participant's pain intensity. The participant indicates their level of pain on average and at its worst during work or at rest over the past 3 days.
Range of motion of the neck | 8 weeks
  The range of motion of the neck is measured by using motion capture system with the IMU (inertial measurement unit) sensors.
Pain pressure threshold (kg/m2) | 8 weeks
  The pain pressure threshold is measured by using a hand-held dynamometer.
Neck disability index (NDI, 0~100%) | 8 weeks
  The NDI is a questionnaire used for assessing self-rated disability in patient participant with neck pain of mechanical origin.
Beck Anxiety Inventory (BAI, scoring from 0~63) | 8 weeks
  The BAI is a brief, self-report assessment for measuring anxiety severity and level.

CONTACTS AND LOCATIONS:
Locations (1):
- WanFang Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No